CLINICAL TRIAL: NCT06001294
Title: The Value of Serum ELABELA in Early Diagnosis of Sepsis-Associated Acute Kidney Injury
Brief Title: We Collected Blood Samples From Septic Shock Patients and Measured ELABELA, Creatinine, and NGAL Levels. Survival After 7 Days Was Recorded and Analyzed to Evaluate the Potential of Serum ELABELA as an Early Diagnostic Marker for Sepsis-associated Acute Kidney Injury.
Acronym: ELABELA（ELA）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangcheng Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiangcheng Zhang, Director of Intensive Care Medicine Department, Huai'an First People's Hospital, Huai'an No.1 People's Hospital
Organization: Huai'an No.1 People's Hospital (Other)
Other Study IDs: Huaian1H
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: sepsis associated acute kidney injury; ELABELA
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators selected patients diagnosed with sepsis who were admitted to the Intensive Care Unit (ICU) of Huai'an First People's Hospital between June 2022 and December 2023, as well as healthy individuals with normal kidney function during the same period, for the research. The investigators collected blood samples from patients with septic shock or sepsis at 6 hours, 12 hours, 24 hours, 48 hours, 3 days, 5 days, and 7 days after diagnosis， and also collected blood samples from the healthy individuals. The blood samples were stored in gel separation vacuum tubes containing heparin as an anticoagulant. The supernatant was removed and stored at -80°C, and the levels of plasma ELA (enzyme-linked immunosorbent assay) were measured using a standardized ELA kit. Additionally, serum NGAL (neutrophil gelatinase-associated lipocalin) and creatinine levels were measured simultaneously. The subjects were divided into three groups based on the KDIGO diagnostic criteria: sepsis-associated acute kidney injury (S-AKI) group, sepsis non-AKI group, and normal control group. Finally, the data were analyzed to determine the early diagnostic value of ELA for S-AKI. Approximately 70 specimens were collected in total.

ELIGIBILITY:
Inclusion Criteria:

Patients with sepsis admitted to the ICU.

Exclusion Criteria:

1. Under 18 years old;
2. History of chronic kidney disease;
3. Recipients of organ transplantation within the past year;
4. Patients or their families could not give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-07-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The value of ELABELA | Venous blood samples were collected at 6 hours, 12 hours, 24 hours, 48 hours, 3 days, 5 days and 7 days after the diagnosis of sepsis or septic shock
  Significance of serum ELABELA in the early diagnosis of sepsis-associated renal injury.

SECONDARY OUTCOMES:
7-day survival rate | 7-day
  The significance of serum ELABELA in evaluating the short-term prognosis of sepsis-associated renal injury.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Zhang, Study Director — Huai'an No.1 People's Hospital
Locations (1):
- Department of Critical Care Medicine, The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huaian, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Section 2: AKI Definition. Kidney Int Suppl (2011). 2012 Mar;2(1):19-36. doi: 10.1038/kisup.2011.32. No abstract available. PMID 25018918
- [Background] Ronco C, Bellomo R, Kellum JA. Acute kidney injury. Lancet. 2019 Nov 23;394(10212):1949-1964. doi: 10.1016/S0140-6736(19)32563-2. PMID 31777389
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Bagshaw SM, Lapinsky S, Dial S, Arabi Y, Dodek P, Wood G, Ellis P, Guzman J, Marshall J, Parrillo JE, Skrobik Y, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Acute kidney injury in septic shock: clinical outcomes and impact of duration of hypotension prior to initiation of antimicrobial therapy. Intensive Care Med. 2009 May;35(5):871-81. doi: 10.1007/s00134-008-1367-2. Epub 2008 Dec 9. PMID 19066848
- [Background] Bagshaw SM, Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten HM, Ronco C, Kellum JA; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Septic acute kidney injury in critically ill patients: clinical characteristics and outcomes. Clin J Am Soc Nephrol. 2007 May;2(3):431-9. doi: 10.2215/CJN.03681106. Epub 2007 Mar 21. PMID 17699448
- [Background] Wen Y, Parikh CR. Current concepts and advances in biomarkers of acute kidney injury. Crit Rev Clin Lab Sci. 2021 Aug;58(5):354-368. doi: 10.1080/10408363.2021.1879000. Epub 2021 Feb 8. PMID 33556265
- [Background] Chng SC, Ho L, Tian J, Reversade B. ELABELA: a hormone essential for heart development signals via the apelin receptor. Dev Cell. 2013 Dec 23;27(6):672-80. doi: 10.1016/j.devcel.2013.11.002. Epub 2013 Dec 5. PMID 24316148
- [Background] Chen H, Wang L, Wang W, Cheng C, Zhang Y, Zhou Y, Wang C, Miao X, Wang J, Wang C, Li J, Zheng L, Huang K. ELABELA and an ELABELA Fragment Protect against AKI. J Am Soc Nephrol. 2017 Sep;28(9):2694-2707. doi: 10.1681/ASN.2016111210. Epub 2017 Jun 5. PMID 28583915